CLINICAL TRIAL: NCT00610623
Title: Proof of Concept Study to Investigate the Impact of Azithromycin Administered iv Versus Placebo on the Prevention of Pneumonia in Ventilated Patients Colonized by Pseudomonas Aeruginosa
Brief Title: Azithromycin as a Quorum-Sensing Inhibitor for the Prevention of Pseudomonas Aeruginosa Ventilator-Associated Pneumonia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The sponsor decided to stop the study prematurely because of financial issues
Sponsor: Anbics Management-Services Ag (Industry)
Collaborators: Swiss National Science Foundation (Other)
Responsible Party: Christian van Delden, Service of Infectious Diseases, University Hospital Geneva
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Anb006#2001
Record Dates: First submitted 2008-01-24; First posted 2008-02-08 (Estimated); Last update posted 2008-02-08 (Estimated); Status verified 2008-01

CONDITIONS: Pneumonia, Ventilator-Associated; Pseudomonas Infections
Keywords: Pseudomonas aeruginosa; Pneumonia; Ventilator-Associated; Quorum Sensing
MeSH Terms: conditions — Pneumonia, Ventilator-Associated; Pseudomonas Infections; Pneumonia | interventions — Azithromycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): azithromycin iv 300 mg/day
  Interventions: Drug: azithromycin
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: azithromycin — 300 mg/day, IV from day 1 to 20
  Other Names: Zithromax
  Arms: 1
Drug: placebo — once per day, IV from day 1 to 20
  Arms: 2

SUMMARY:
The purpose of this study is to assess the clinical efficacy of azithromycin, used as a quorum-sensing blocker, when compared to placebo for preventing or delaying the occurrence of pneumonia in ventilated patients colonized with Pseudomonas aeruginosa.

ELIGIBILITY:
Inclusion Criteria:

* Male and non pregnant female aged 18 to 75 years
* Patients hospitalized in ICU, under mechanically assisted ventilation expected to be mandatory for 3 days or more
* Reasonable survival chance within next few days with an Apache score 10-25
* Tracheal aspirate found positive for P. aeruginosa
* The subject (or a close family member in case of incompetence) understands the procedure, agrees to participate, and is willing to give written informed consent
* Informed consent must be obtained for all subjects before enrollment in the study, by patient or by a close family member

Exclusion Criteria:

* Poor prognosis as judged by Apache score II score >25
* Pregnant female
* Grossly under-or overweight (BMI<18or >29)
* Ongoing therapy with a macrolide
* Known allergy to any macrolide
* Proven P. aeruginosa pneumonia
* Ongoing anti-pseudomonal therapy with a proven susceptible colonizing strain
* Anticipated short duration of mechanical ventilation (<3 days)
* Known drug interaction that could either decrease efficacy or raise safety concerns
* Severe hepatic failure (type C, score >10 on Child Pugh scale)
* Sick sinus syndrome or long QT syndrome
* Recent donation of blood or participation in another clinical trial within 3 months
* Any situation exposing the patient to higher risk or possibly confounding results

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2003-04; Primary Completion 2005-10 (Actual); Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
Occurrence of and time to Pseudomonas aeruginosa pneumonia | daily

SECONDARY OUTCOMES:
occurrence of and time to death | daily
time to extubation | daily
overall outcome | daily
duration of hospitalization and ICU stay | daily
occurrence of infections to other bacterial strains | daily
cost assessment | daily
demonstrate using in vitro and in vivo parameters that azithromycin can be used as a quorum-sensing blocker against P. aeruginosa | daily
determine whether prolonged treatment with azithromycin may induce resistance to any of 11 anti-pseudomonal antibiotics | daily
determine whether P. aeruginosa can develop resistance to the quorum-sensing effect of azithromycin | daily

CONTACTS AND LOCATIONS:
Overall Officials: Christian Van Delden, MD, Principal Investigator — Service of Infectious Diseases, University Hospital Geneva, Switzerland; Jean Carlet, MD, Study Chair — General Intensive Care Unit, Hospital Saint-Joseph, Paris, France
Locations (20):
- Belgium (2):
  - General Intensive Car Unit, Centre Hospitalier Universitaire de Liège, Liège, Liège
  - Intensive Care Unit, Clinique Saint-Pierre, Ottignies, Louvain
- France (8):
  - Intensive Care Unit, Jean Minjoz University Hospital, Besançon, Besancon
  - Intensive Car Unit, Calmette University Hospital of Lille, Lille, Lille
  - Medical-surgical intensive car unit, Dupuytren Teaching Hospital, Limoges, Limoges
  - General Intensive Care Unit, Montauban City Hospital, Montauban, Montauban
  - Medical Intensive Car Unit, Hospital Bichat, Paris, Paris
  - Surgical Intensive Car Unit; University Hospital Bichat, Paris, Paris
  - General Intensive Care Unit, Hospital Saint-Joseph, Paris, Paris
  - Medical Intensive Care Unit, Cochin Hospital, Paris, Paris
- Poland (3):
  - Intensive Care Unit, Wojewodzki Hospital, Krakow
  - Intensive Care Unit, Wojewodzki Hospital, Sosnowiec
  - Intensive Care Unit, Central Hospital, Warsaw
- Serbia and Montenegro (2):
  - Surgical Intensive Care Unit, Clinical Center of Serbia, Institut of Neurosurgery, Belgrade
  - Surgical Intensive Care Unit, Clinical Center of Serbia, Belgrade
- Spain (4):
  - Intensive Care Unit, Hospital del Mar, Barcelona, Barcelona
  - Internal Medicine, Vall d'Hebron Hospital, Barcelona, Barcelona
  - Intensive Care Unit, Joan XXIII University Hospital, Tarragona, Tarragona
  - Intensive Care Unit, San Dureta University Hospital, Palma de Mallorca
- Surgical and Medical Intensive Care Units, University Hospital Lausanne, Lausanne, Canton of Vaud, Switzerland

REFERENCES:
- [Derived] Kohler T, Perron GG, Buckling A, van Delden C. Quorum sensing inhibition selects for virulence and cooperation in Pseudomonas aeruginosa. PLoS Pathog. 2010 May 6;6(5):e1000883. doi: 10.1371/journal.ppat.1000883. PMID 20463812